CLINICAL TRIAL: NCT04791514
Title: An Open-Label Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Treprostinil Palmitil Inhalation Powder in Participants With Pulmonary Arterial Hypertension
Brief Title: A Study of Treprostinil Palmitil Inhalation Powder (TPIP) In Pulmonary Arterial Hypertension (PAH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrolment
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INS1009-201
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Treprostinil Palmitil Inhalation Powder; Treprostinil Palmitil
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treprostinil Palmitil Inhalation Powder (Experimental): Participant received a single dose of TPIP 112.5 micrograms (μg) via oral inhalation on Day 1. The participant then entered into a 16-week Extended Use Treatment (EUT) Period during which TPIP, administered via oral inhalation, was titrated up to a mean daily dose of 320 μg.
  Interventions: Drug: Treprostinil Palmitil

INTERVENTIONS:
Drug: Treprostinil Palmitil — Administered by oral inhalation using a Plastiape capsule-based dry powder inhaler
  Other Names: INS1009

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of single dose of treprostinil palmitil inhalation powder (TPIP) in participants with pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age at the time of signing the informed consent
* Participants must have a diagnosis of World Health Organization Group 1 Pulmonary Hypertension (PH) (PAH) with the following characteristics

  1. Etiology of idiopathic, heritable, drug/toxin-induced or connective tissue disease (CTD)-related PAH
  2. Right heart catheterization with the following hemodynamic findings:
* Mean pulmonary arterial pressure (mPAP) > 20 mmHg at rest,
* Pulmonary capillary wedge pressure (PCWP) ≤ 15 mmHg, and
* Pulmonary vascular resistance (PVR) of ≥ 3 Wood Units (WU)
* No change in pulmonary hypertension medications (eg, ambrisentan, bosentan, macitentan, sildenafil, tadalafil, riociguat) or dosage for at least 90 days prior to Screening
* No change in diuretic use or dosage for at least 30 days prior to Screening
* Body mass index (BMI) within the range 18.0 - 32.0 kg/m^2 (inclusive)
* Male participants: Male participants and their female partners of childbearing potential must agree to use highly effective contraception from Study Day 1 to at least 90 days after dosing
* Female participants: Women of child-bearing potential (WOCPB, defined as premenopausal, not surgically sterile for at least 3 months prior to Screening) must use a highly effective contraception method and agree to be tested for pregnancy from at Screening, Baseline, and 30 days after dosing
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.

Exclusion Criteria:

* Any PH other than idiopathic, hereditary, drug/toxin-induced, or connective tissue disease (CTD) associated PAH (eg, congenital heart disease-associated PAH, portal hypertension-associated PAH, PH belonging to Groups 2 through 5)
* Allergy, or documented hypersensitivity or contraindication, to the ingredients of treprostinil palmitil inhalation powder (TPIP) or treprostinil (TRE)
* Previous intolerance to prostacyclin analogs or receptor agonists (eg, selexipag) per investigator discretion
* History of anaphylaxis or previously documented hypersensitivity reaction to any drug per Investigator discretion
* History of heart disease including left ventricular ejection fraction (LVEF) ≤ 40% or clinically significant valvular, constrictive, or atherosclerotic heart disease (myocardial infarction, etc)
* Active liver disease or hepatic dysfunction manifested as:

  1. Elevated liver function test results (ALT or AST > 2 × ULN) at Screening
  2. Bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN; ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) at Screening.
  3. Known hepatic or biliary abnormalities, not including Gilbert's syndrome or asymptomatic gallstones at Screening.
* History of HIV infection/positive HIV serology test result at Screening
* History of active/chronic Hepatitis B or C/ positive hepatitis B or C serology test result at Screening
* History of abnormal bleeding or bruising
* Known or suspected immunodeficiency disorder, including history of invasive opportunistic infections (eg, tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution, or otherwise recurrent infections of abnormal frequency, or prolonged infections suggesting an immune-compromised status, as judged by the investigator
* Active and current symptomatic infection by SARS CoV 2
* Participants with current or recent (past 4 weeks) lower respiratory tract infection
* History of malignancy in the past 5 years, with exception of completely treated in situ carcinoma of the cervix and completely treated non-metastatic squamous or basal cell carcinoma of the skin
* Participants receiving triple combination therapy for PAH consisting of endothelin receptor agonists, phosphoesterase type 5 inhibitors, and guanylate cyclase stimulators (riociguat)
* Participants receiving prostanoids/prostacyclin agonists
* Participants receiving potent CYP2C8 inhibitors, such as gemfibrozil
* Have participated in any other interventional clinical studies within 30 days of Baseline
* Current or history of substance and/or alcohol abuse
* Current user of cigarettes or e-cigarettes
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- USA002, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated by the Sponsor due to low enrolment. As only 1 participant was enrolled in this study, no data is reported here, in order to protect and maintain participant privacy/confidentiality.
Groups:
- Treprostinil Palmitil Inhalation Powder (TPIP): Participant received a single dose of TPIP 112.5 micrograms (μg) via oral inhalation on Day 1. The participant then entered into a 16-week Extended Use Treatment (EUT) Period during which TPIP, administered via oral inhalation, was titrated up to a mean daily dose of 320 μg.
Period: Overall Study
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor due to low enrolment. As only 1 participant was enrolled in this study, no data is reported here, in order to protect and maintain participant privacy/confidentiality.
Groups:
- Treprostinil Palmitil Inhalation Powder (TPIP): Participant received a single dose of TPIP 112.5 μg via oral inhalation on Day 1. The participant then entered into a 16-week EUT Period during which TPIP, administered via oral inhalation, was titrated up to a mean daily dose of 320 μg.
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex/Gender, Customized
Race/Ethnicity, Customized
Race/Ethnicity, Customized

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience a Treatment Emergent Adverse Event (TEAE)
Time Frame: Up to 150 days
Population: as for baseline characteristics
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) After TPIP Administration
Time Frame: Day 1: Pre-treatment (Baseline), 8 and 24 hours post-treatment
Population: as for baseline characteristics
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Number analyzed (Participants) | 0

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of Treprostinil (TRE) in Plasma
Time Frame: Pre-dose and multiple timepoints post-dose up to Day 2
Population: as for baseline characteristics
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Maximum Concentration (Tmax) of Treprostinil (TRE) in Plasma
Time Frame: Pre-dose and multiple timepoints post-dose up to Day 2
Population: as for baseline characteristics
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Number analyzed (Participants) | 0

5. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time of the Last Measurable Concentration (AUClast) of Treprostinil (TRE) in Plasma
Time Frame: Pre-dose and multiple timepoints post-dose up to Day 2
Population: as for baseline characteristics
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Number analyzed (Participants) | 0

6. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-∞) of Treprostinil (TRE) in Pasma
Time Frame: Pre-dose and multiple timepoints post-dose up to Day 2
Population: as for baseline characteristics
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Number analyzed (Participants) | 0

7. Secondary Outcome: Elimination Half-life (t1/2) of Treprostinil (TRE) in Plasma
Time Frame: Pre-dose and multiple timepoints post-dose up to Day 2
Population: as for baseline characteristics
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 150 days
Description: The study was terminated by the Sponsor due to low enrolment. As only 1 participant was enrolled in this study, no data is reported here, in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Treprostinil Palmitil Inhalation Powder (TPIP)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor due to low enrolment. As only 1 participant was enrolled in this study, no data is reported here, in order to protect and maintain participant privacy/confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT04791514/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT04791514/SAP_001.pdf